CLINICAL TRIAL: NCT06784739
Title: COMMUNITY - the COVID-19 Immunity Study
Acronym: COMMUNITY
Status: Recruiting | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Thålin, MD, PhD, Karolinska Institutet
Other Study IDs: 2020-01653; 2020-01653 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2025-01-16; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: COVID 19; Respiratory Synctial Virus; Influenza Virus; SARS-CoV-2 Virus
Keywords: COVID-19; Mucosal immunity; Pandemic; Vaccination; Secretory IgA
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, PBMC, saliva, nasal secretions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The COMMUNITY cohort - healthcare workers: 5000 healthcare workers employed at Danderyd Hospital at time of enrollment
  Interventions: Other: Blood sampling; Other: Mucosal sampling; Diagnostic Test: PCR-test
- The COMMUNITY cohort - COVID-19 patients: 500 patients admitted to Danderyd Hospital with confirmed SARS-CoV-2 infection
  Interventions: Other: Blood sampling; Other: Mucosal sampling; Diagnostic Test: PCR-test

INTERVENTIONS:
Other: Blood sampling — Venous blood sampling
Other: Mucosal sampling — Saliva and nasal secretions
Diagnostic Test: PCR-test — RT qPCR test to determine infection with SARS-CoV-2, Influenza A/B and/or RSV A/B.

SUMMARY:
The principal aim of the COMMUNITY study is to investigate immune responses following SARS-CoV-2 infection and/or vaccination in healthcare workers and hospitalized COVID-19 patients. The study aims to enroll a total of 5,000 healthcare workers and 500 COVID-19 patients. All participants are enrolled at Danderyd Hospital in Stockholm, Sweden. Participants will be followed every four months with blood and mucosal sampling in addition to demographic and clinical data provided by the participants and from national registries.

Primary outcome:

- Antibody responses in blood and mucosa following SARS-CoV-2 infection and/or vaccination

Secondary outcomes:

* Cellular immune responses following SARS-CoV-2 infection and/or vaccination
* Antibody responses in blood and mucosa following following Influenza A/B infection and/or vaccination
* Antibody responses in blood and mucosa following following RSV A/B infection

Blood and mucosal samples are collected every 4 months and at tighter intervals in sub studies. PCR testing is conducted upon symptoms of respiratory infections and with regular intervals regardless of symptomatology in sub studies. Participants provide detailed demographic and clinical data through a smart phone application-based questionnaire. Data on infection and vaccination history is collected from national registries

DETAILED DESCRIPTION:
The COMMUNITY study is designed to longitudinally follow healthcare workers and recovered COVID-19 patients to assess SARS-CoV-2 immune responses over time. Follow-ups are conducted every four months, including serum, PBMC, and mucosa (saliva and nasal secretions) samples. Sub studies with additional samplings and PCR screenings are conducted with regular intervals to assess vaccine responses and correlates to protection against infection.

Analyses include:

* Quantification and characterization of antibody responses
* Evaluation of T and B-cell responses
* RT-qPCR detection of viral infection
* Mucosal microbiome evaluation

Clinical and demographic data, including information on hospital workplace, exposure, immunosuppressive treatments or conditions, and results from SARS-CoV-2 Rapid Diagnostic Tests, are collected at each follow-up through a smartphone-based app system. Data on SARS-CoV-2 infections and vaccinations are obtained from national registries. In addition, data from home based PCR-screenings are continuously being monitored for SARS-CoV-2, Influenza and RSV infections.

All samples are stored in Biobank Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Health care workers: Employment at Danderyd hospital at time of enrollment
* COVID-19 patients: Admitted to Danderyd Hospital with confirmed SARS-CoV-2 infection at time of enrollment

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danderyd Hospital employs approximately 4,500 healthcare workers. All HCWs are invited to participate in the study through information disseminated via the hospital intranet, email, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Antibody responses following SARS-CoV-2 infection and/or vaccination | 2022-2026
  Antigen-specific IgG and IgA responses in serum, saliva and nasal secretions (trajectories over time and correlates to protection against infection)

SECONDARY OUTCOMES:
Antibody responses following Influenza A/B infection and/or vaccination | 2022-2026
  Antigen-specific IgG and IgA responses in serum, saliva and nasal secretions (trajectories over time and correlates to protection against infection)
Antibody responses following RSV infection | 2020-2026
  Antigen-specific IgG and IgA responses in serum, saliva and nasal secretions (trajectories over time and correlates to protection against infection)
Cellular immune responses following SARS-CoV-2, Influenza A/B and RSV A/B infection and/or vaccination | 2020-2026
  T and B cell responses in blood

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Thålin, MD, PhD, Principal Investigator — Department of Clinical Sciences, Karolinska Institutet Danderyd Hospital
Locations (2):
- Sweden (2):
  - Danderyd hospital, Stockholm
  - Karolinska Institutet Danderyd Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Under consideration

REFERENCES:
- [Background] Ng H, Havervall S, Rosell A, Aguilera K, Parv K, von Meijenfeldt FA, Lisman T, Mackman N, Thalin C, Phillipson M. Circulating Markers of Neutrophil Extracellular Traps Are of Prognostic Value in Patients With COVID-19. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):988-994. doi: 10.1161/ATVBAHA.120.315267. Epub 2020 Dec 3. PMID 33267662
- [Background] Sachetto ATA, Archibald SJ, Hisada Y, Rosell A, Havervall S, van Es N, Nieuwland R, Campbell RA, Middleton EA, Rondina MT, Thalin C, Mackman N. Tissue factor activity of small and large extracellular vesicles in different diseases. Res Pract Thromb Haemost. 2023 Mar;7(3):100124. doi: 10.1016/j.rpth.2023.100124. Epub 2023 Mar 15. PMID 37012986
- [Background] Monteil V, Eaton B, Postnikova E, Murphy M, Braunsfeld B, Crozier I, Kricek F, Niederhofer J, Schwarzbock A, Breid H, Devignot S, Klingstrom J, Thalin C, Kellner MJ, Christ W, Havervall S, Mereiter S, Knapp S, Sanchez Jimenez A, Bugajska-Schretter A, Dohnal A, Ruf C, Gugenberger R, Hagelkruys A, Montserrat N, Kozieradzki I, Hasan Ali O, Stadlmann J, Holbrook MR, Schmaljohn C, Oostenbrink C, Shoemaker RH, Mirazimi A, Wirnsberger G, Penninger JM. Clinical grade ACE2 as a universal agent to block SARS-CoV-2 variants. EMBO Mol Med. 2022 Aug 8;14(8):e15230. doi: 10.15252/emmm.202115230. Epub 2022 Jul 4. PMID 35781796
- [Background] Mravinacova S, Jonsson M, Christ W, Klingstrom J, Yousef J, Hellstrom C, Hedhammar M, Havervall S, Thalin C, Pin E, Tegel H, Nilsson P, Manberg A, Hober S. A cell-free high throughput assay for assessment of SARS-CoV-2 neutralizing antibodies. N Biotechnol. 2022 Jan 25;66:46-52. doi: 10.1016/j.nbt.2021.10.002. Epub 2021 Oct 7. PMID 34628049
- [Result] Havervall S, Jernbom Falk A, Klingstrom J, Ng H, Greilert-Norin N, Gabrielsson L, Salomonsson AC, Isaksson E, Rudberg AS, Hellstrom C, Andersson E, Olofsson J, Skoglund L, Yousef J, Pin E, Christ W, Olausson M, Hedhammar M, Tegel H, Mangsbo S, Phillipson M, Manberg A, Hober S, Nilsson P, Thalin C. SARS-CoV-2 induces a durable and antigen specific humoral immunity after asymptomatic to mild COVID-19 infection. PLoS One. 2022 Jan 12;17(1):e0262169. doi: 10.1371/journal.pone.0262169. eCollection 2022. PMID 35020778
- [Result] von Meijenfeldt FA, Havervall S, Adelmeijer J, Thalin C, Lisman T. Persistent endotheliopathy in the pathogenesis of long COVID syndrome: Comment from von Meijenfeldt et al. J Thromb Haemost. 2022 Jan;20(1):267-269. doi: 10.1111/jth.15580. Epub 2021 Nov 22. No abstract available. PMID 34731533
- [Result] Blom K, Bladh O, Havervall S, Marking U, Greilert Norin N, Alm JJ, Klingstrom J, Thalin C. Point prevalence of SARS-CoV-2 infection among healthcare workers in March and June 2023 in Sweden. Lancet Reg Health Eur. 2023 Aug 30;33:100725. doi: 10.1016/j.lanepe.2023.100725. eCollection 2023 Oct. No abstract available. PMID 37680234
- [Result] von Meijenfeldt FA, Havervall S, Adelmeijer J, Lundstrom A, Magnusson M, Mackman N, Thalin C, Lisman T. Sustained prothrombotic changes in COVID-19 patients 4 months after hospital discharge. Blood Adv. 2021 Feb 9;5(3):756-759. doi: 10.1182/bloodadvances.2020003968. No abstract available. PMID 33560386
- [Result] Havervall S, Rosell A, Phillipson M, Mangsbo SM, Nilsson P, Hober S, Thalin C. Symptoms and Functional Impairment Assessed 8 Months After Mild COVID-19 Among Health Care Workers. JAMA. 2021 May 18;325(19):2015-2016. doi: 10.1001/jama.2021.5612. PMID 33825846
- [Result] Blom K, Marking U, Havervall S, Norin NG, Gordon M, Garcia M, Tecleab T, Christ W, Forsell M, Phillipson M, Nilsson P, Mangsbo S, Hober S, Aberg M, Klingstrom J, Thalin C. Immune responses after omicron infection in triple-vaccinated health-care workers with and without previous SARS-CoV-2 infection. Lancet Infect Dis. 2022 Jul;22(7):943-945. doi: 10.1016/S1473-3099(22)00362-0. Epub 2022 Jun 9. No abstract available. PMID 35691303
- [Result] Havervall S, Marking U, Greilert-Norin N, Gordon M, Ng H, Christ W, Phillipson M, Nilsson P, Hober S, Blom K, Klingstrom J, Mangsbo S, Aberg M, Thalin C. Impact of SARS-CoV-2 infection on vaccine-induced immune responses over time. Clin Transl Immunology. 2022 Apr 18;11(4):e1388. doi: 10.1002/cti2.1388. eCollection 2022. PMID 35444806
- [Result] von Meijenfeldt FA, Havervall S, Adelmeijer J, Lundstrom A, Magnusson M, Mackman N, Thalin C, Lisman T. COVID-19 is Associated with an Acquired Factor XIII Deficiency. Thromb Haemost. 2021 Dec;121(12):1668-1669. doi: 10.1055/a-1450-8414. Epub 2021 May 5. No abstract available. PMID 33742434
- [Result] Blom K, Havervall S, Marking U, Norin NG, Bacchus P, Groenheit R, Brave A, Thalin C, Klingstrom J. Infection Rate of SARS-CoV-2 in Asymptomatic Healthcare Workers, Sweden, June 2022. Emerg Infect Dis. 2022 Oct;28(10):2119-2121. doi: 10.3201/eid2810.221093. Epub 2022 Aug 23. PMID 35997692
- [Result] Bladh O, Aguilera K, Marking U, Kihlgren M, Greilert Norin N, Smed-Sorensen A, Sallberg Chen M, Klingstrom J, Blom K, Russell MW, Havervall S, Thalin C, Aberg M. Comparison of SARS-CoV-2 spike-specific IgA and IgG in nasal secretions, saliva and serum. Front Immunol. 2024 Mar 15;15:1346749. doi: 10.3389/fimmu.2024.1346749. eCollection 2024. PMID 38558811
- [Result] Bladh O, Marking U, Havervall S, Norin NG, Aguilera K, Hober S, Smed-Sorensen A, Gordon M, Blom K, Aberg M, Klingstrom J, Thalin C. Mucosal immune responses following a fourth SARS-CoV-2 vaccine dose. Lancet Microbe. 2023 Jul;4(7):e488. doi: 10.1016/S2666-5247(23)00102-7. Epub 2023 Apr 20. No abstract available. PMID 37086736
- [Result] Marking U, Bladh O, Havervall S, Greilert-Norin N, Gordon M, Alm JJ, Blom K, Aberg M, Klingstrom J, Thalin C. Mucosal IgA protects against BQ.1 and BQ.1.1 infection. Lancet Infect Dis. 2023 Aug;23(8):e272-e273. doi: 10.1016/S1473-3099(23)00421-8. Epub 2023 Jul 12. No abstract available. PMID 37453441
- [Result] Havervall S, Marking U, Svensson J, Greilert-Norin N, Bacchus P, Nilsson P, Hober S, Gordon M, Blom K, Klingstrom J, Aberg M, Smed-Sorensen A, Thalin C. Anti-Spike Mucosal IgA Protection against SARS-CoV-2 Omicron Infection. N Engl J Med. 2022 Oct 6;387(14):1333-1336. doi: 10.1056/NEJMc2209651. Epub 2022 Sep 14. No abstract available. PMID 36103621
- [Result] Marking U, Bladh O, Aguilera K, Yang Y, Greilert Norin N, Blom K, Hober S, Klingstrom J, Havervall S, Aberg M, Sheward DJ, Thalin C. Humoral immune responses to the monovalent XBB.1.5-adapted BNT162b2 mRNA booster in Sweden. Lancet Infect Dis. 2024 Feb;24(2):e80-e81. doi: 10.1016/S1473-3099(23)00779-X. Epub 2024 Jan 5. No abstract available. PMID 38190833
- [Result] Bladh O, Greilert-Norin N, Havervall S, Marking U, Aguilera K, Alm JJ, Blom K, Aberg M, Klingstrom J, Thalin C. Mucosal and Serum Antibodies 3 Weeks after Symptomatic BA.2.86 Infection. N Engl J Med. 2023 Oct 26;389(17):1626-1628. doi: 10.1056/NEJMc2310347. No abstract available. PMID 37888924
- See also: Charlotte Thålin Group at KI — https://ki.se/en/research/research-areas-centres-and-networks/research-groups/medicine-at-ki-ds